CLINICAL TRIAL: NCT02364297
Title: Efficacy of Early-TIPS in the Treatment of Acute Variceal Bleeding From Gastric Fundal Varices: a RCT vs Standard Therapy
Brief Title: TIPS in Fundal Variceal Bleeding (the TFB Study)
Acronym: TFB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitario Ramon y Cajal (Other); Hospital del Mar (Other)
Responsible Party: Principal Investigator, Àngels Escorsell, Senior Consultant, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET_GV15; PI 14/00392 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Portal Hypertension; Bleeding Gastric Varices
Keywords: Bleeding gastric varices; Transjugular intrahepatic portosystemic shunt (TIPS); Injection of adhesives
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early TIPS (Active Comparator): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic injection of tissue adhesives according to the center protocol.
  Performance of TIPS in the first 5 days following acute gastric variceal bleeding.
  Interventions: Device: Early TIPS
- Control (Placebo Comparator): Standard treatment to achieve initial hemostasis: vasoactive drugs (somatostatin or terlipressin) + endoscopic injection of tissue adhesives according to the center protocol.
  Standard combined endoscopic and pharmacological therapy as a secondary prophylaxis (beta-blockers or carvedilol + repeated injection of tissue adhesives until the erradication of the fundal varices).
  Interventions: Device: Early TIPS

INTERVENTIONS:
Device: Early TIPS — TIPS (first 5 days)

SUMMARY:
In the last years, important advances have been done in the treatment and prevention of fundal variceal bleeding in patients with cirrhosis. Experts agree that the combination of pharmacological and endoscopic therapy (with tissue adhesives) should be the first line therapy in the acute bleeding episode from isolated gastric varices (IGV1) or type 2 gastroesophageal varices (GOV2) varices; whereas transjugular intrahepatic portosystemic shunt (TIPS) is considered a rescue therapy. TIPS has been shown to effectively prevent variceal rebleeding but with a potential increase in the incidence of hepatic encephalopathy and/or liver failure. In this sense, a recent randomized controlled trial (RCT) in esophageal variceal bleeding showed that an early TIPS, performed during the first 72h after patient admission resulted in a significant decrease in failure to control bleeding and early and late rebleeding. Moreover, survival was also significantly increased as well as other portal-hypertension related complications (ascites, spontaneous bacterial peritonitis, hepatorenal syndrome, etc).

The present study is directed at comparing the outcome of patients with acute bleeding from fundal varices (IGV1 or GOV2) treated by standard therapy (vasoactive drugs + endoscopic injection of tissue adhesives) with or without early TIPS (performed during the first 1-5 days after admission). Main end-point will be survival free of variceal rebleeding at 1 year from inclusion.

ELIGIBILITY:
Inclusion Criteria:

Patients developing acute variceal bleeding from GOV2 and/or IGV1 defined according to Baveno II criteria, admitted in the Hospital and receiving standard combined medical therapy (somatostatin 3 mg/12h continuous IV infusion or terlipressin, 2mg/4h IV + endoscopic injection of tissue adhesives as per center protocol).

Exclusion Criteria:

* Hepatocarcinoma without therapeutic options (according to Milan criteria).
* Portal or mesenteric vein thrombosis avoiding the performance of TIPS.
* Acute alcoholic hepatitis.
* Platelet count < 20.000/mm3.
* Previous treatment with portosystemic shunt.
* Pregnancy.
* Previous inclusion in the current study.
* Terminal liver disease (bilirrubin > 10 mg/dL and/or prothrombin index < 30%); or other fatal non-liver diseases.
* Denied informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Combined: Absence of rebleeding + survival | 1 year
  The primary endpoint combines absence of rebleeding + survival during the first 1 year after inclusion in the study. Patients to compare are those with liver cirrhosis and acute bleeding from IGV1 or GOV2 varices initially treated with combined pharmacological and endoscopic therapy. Those patients will be randomized to receive a TIPS or standard medical therapy (pharmacological + endoscopic injection of tissue adhesives)

SECONDARY OUTCOMES:
Absence of portal hypertension-related complications (ascites, spontaneous bacterial peritonitis, hepatorenal syndrome) | 6 weeks and 1 year
  Comparison of the development of portal-hypertension related complications.
Transfusional requirements | 6 weeks and 1 year
  We will compare the number of packed red blood cells required by each treatment arms as a surrogate of rebleeding.
Individual adverse events | 1 year
  Related and not related to the therapies under study.
Hospital stay | 1 year
  Including the stay for the index bleed and also readmissions due to complications of liver disease.
Use of hospital resources | 1 year
  Use of hospital resources other than specified in the treatment arms (TIPS, revision of TIPS patency, derivative surgery or additional endoscopic therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Angels Escorsell, MD, Principal Investigator — Senior Consultant. Liver Unit
Locations (5):
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona, Catalonia
  - ICU Liver Unit. Hospital Clinic of Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Arnau de Vilanova, Lleida

REFERENCES:
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Background] Garcia-Tsao G, Bosch J, Groszmann RJ. Portal hypertension and variceal bleeding--unresolved issues. Summary of an American Association for the study of liver diseases and European Association for the study of the liver single-topic conference. Hepatology. 2008 May;47(5):1764-72. doi: 10.1002/hep.22273. No abstract available. PMID 18435460
- [Result] Garcia-Pagan JC, Caca K, Bureau C, Laleman W, Appenrodt B, Luca A, Abraldes JG, Nevens F, Vinel JP, Mossner J, Bosch J; Early TIPS (Transjugular Intrahepatic Portosystemic Shunt) Cooperative Study Group. Early use of TIPS in patients with cirrhosis and variceal bleeding. N Engl J Med. 2010 Jun 24;362(25):2370-9. doi: 10.1056/NEJMoa0910102. PMID 20573925